CLINICAL TRIAL: NCT05837104
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Assess the Efficacy and Safety of Magnesium Vitamin B6 in Combination With Treatment as Usual in First Episode of Bipolar I Disorder
Brief Title: Efficacy and Safety of Magnesium Vitamin B6 in First Episode Bipolar Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Virginie-Anne Chouinard, MD, Psychiatrist, Psychotic Disorders Division, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022P001911
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Bipolar I Disorder; Depression, Anxiety; Stress
Keywords: First episode Bipolar Disorder; Magnesium vitamin B6; Brain energy metabolism; Depression; Anxiety; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium vitamin B6 (Experimental): Magnesium vitamin B6 (MagnéVie B6®) composed of Magnesium citrate (100mg) and Pyridoxine hydrochloride (10mg) in tablet form, taken three times daily for four weeks.
  Interventions: Drug: Magnesium vitamin B6
- Placebo (Placebo Comparator): Placebo tablet will be taken three times daily for four weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium vitamin B6 — Magnesium citrate (100mg) and Pyridoxine hydrochloride (10mg) in tablet form, taken three times daily for four weeks.
  Other Names: MagnéVie B6®
  Arms: Magnesium vitamin B6
Drug: Placebo — Placebo tablet, three times daily for four weeks.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled proof-of-concept clinical trial to assess the efficacy and safety of Magnesium-vitamin B6in combination with treatment as usual for treating symptoms of depression, stress, and anxiety in patients with first episode bipolar I disorder.

DETAILED DESCRIPTION:
After a first episode of bipolar disorder, subsequent depressive and anxiety symptoms can pose a major challenge to an individual's recovery early in the illness. Individuals often have depressive and anxiety symptoms for a significant proportion of their time. These mood and anxiety symptoms are associated with higher risk for relapse, chronicity and disability. Previous studies have shown that the combination of Magnesium-vitamin B6 has beneficial effects on stress, and depressive and anxiety symptoms. This randomized, double-blind, placebo-controlled trial will assess the benefits of Magnesium-vitamin B6 in combination with treatment as usual (standard of clinical care) on depressive and anxiety symptoms and stress in individuals with bipolar disorder in the early phase of illness. In addition, the investigators aim to assess the effects of Magnesium-vitamin B6 on brain free [Mg2+] and energy metabolism, observed to be altered in bipolar disorder, measured by in vivo 31P magnetic resonance spectroscopy (31P MRS). Magnesium is a promising targeted intervention for bipolar disorder given its significant effects on energy metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Persons between the ages of 18 and 50
* DSM V diagnosis of bipolar I disorder, onset of illness in the last 10 years
* Minimum of two of the following symptoms on the Hamilton Rating Scale of Depression HAM-D (HAM-D, 17 item): depressed mood, feelings of guilt, anxiety-psychic, anxiety-somatic, somatic symptoms-general, somatic symptoms-gastrointestinal.
* Young Mania Rating Scale (YMRS) scores of less than 15
* Ability to sign informed consent.
* Stable disorder and no change in psychiatric medications within 2 weeks of screening and expected to not require addition of any new psychiatric medications during the duration of the 4 weeks of the study.

Exclusion Criteria:

* Unable to sign informed consent.
* Persons weighing over 350lbs.
* Declines to participate.
* Bipolar NOS, Cyclothymia, or Schizoaffective Bipolar type.
* 2 or more manic symptoms that meet DSM-V criteria.
* Persons of childbearing potential who are not using a medically accepted means of contraception.
* Persons who are deemed a serious suicide or homicide risk.
* Unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.
* The following DSM-V diagnoses: 1) substance use disorders, including alcohol, active within 2 months; 2) schizophrenia; 3) delusional disorder; 4) psychotic disorders not otherwise specified; 5) schizoaffective disorder; 6) acute bereavement; 7) severe borderline or antisocial personality disorder.
* Persons meeting criteria for bipolar mixed episode.
* Exposure to levodopa, quinidine, and proton-pump inhibitors within 3 months prior to screening.
* Severe hypomagnesemia (serum magnesium of 0.45 mmol/L).
* Persons who have taken an investigational psychotropic drug within the past 6 months unless the investigational drug was a one-time dose.
* Seizure disorder.
* Dietary supplements including SAMe, St. John's Wort, DHEA, Inositol, and Ginko biloba.
* Previous treatment with the following procedures: vagus nerve stimulation, or deep brain stimulation.
* Have a history of electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) within the last 3 months.
* Have any medical condition that would prevent blood draws.
* Have a history of significant head injury.
* Individuals with galactose intolerance, total lactase deficiency or glucose-galactose malabsorption syndrome (rare hereditary diseases)
* Individuals with allergies to magnesium citrate anhydrous, pyridoxine hydrochloride or any of the other components of Magne B6
* Patients taking psychostimulant medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | 4 weeks
  Change from baseline to week 4 in Hamilton Rating Scale for Depression (HAM-D) total score. Scores range from 0-52; a higher score indicates a higher level of depression.

SECONDARY OUTCOMES:
Change in anxiety symptoms | 4 weeks
  Change from baseline to week 4 in Hamilton Anxiety Rating Scale (HAM-A) total score. Scores range from 0-56; a higher score indicates a higher level of anxiety.
Change in stress symptoms | 4 weeks
  Change from baseline to week 4 in Depression Anxiety Stress Scales (DASS-42) Stress Subscale score. Scores range from 0-42; a higher score indicates a higher level of stress.
Change in Clinical Global Impression (CGI) Scale | 4 weeks
  Change from baseline to week 4 in Clinical Global Impression (CGI) Scale. Scores range from 1-7; a higher score indicates higher severity of illness.
Change in cognitive measure | 4 weeks
  Change from baseline to week 4 in MATRICS Consensus Cognitive Battery (MCCB) Total score. Scores range from 0.00%-100.00%; a higher score indicates higher cognition.
Changes in brain ATP | 4 weeks
  Changes in ATP concentration as measured by in vivo 31P magnetic resonance spectroscopy.
Changes in brain PCr | 4 weeks
  Changes in Phosphocreatine (PCr) concentration as measured by in vivo 31P magnetic resonance spectroscopy.
Changes in brain pH | 4 weeks
  Changes in pH as measured by in vivo 31P magnetic resonance spectroscopy.
Changes in brain inorganic phosphate concentration | 4 weeks
  Changes in inorganic phosphate (Pi) concentration as measured by in vivo 31P magnetic resonance spectroscopy.
Change in brain Mg2+ concentration | 4 weeks
  Change from baseline to week 4 in Mg2+ concentration as measured by 31P MRS.
Change in adverse events | 4 weeks
  Change from baseline to week 4 in adverse events.

OTHER OUTCOMES:
Change in World Health Organization Disability Assessment Schedule (WHODAS) score | 4 weeks
  Change from baseline to week 4 in World Health Organization Disability Assessment Schedule (WHODAS) scale. Scores range from 0-144; a higher score indicates greater dysfunction and disability in major life domains.
Change in World Health Organization Quality of Life (WHOQOL) score | 4 weeks
  Change from baseline to week 4 in World Health Organization Quality of Life (WHOQOL) scale. Scores range from 1-130; a lower score indicates lower perceived quality of life.
Change in Mg blood level | 4 weeks
  Change from baseline to week 4 in Mg blood levels.
Change is Positive and Negative Syndrome Scale (PANSS) total score | 4 weeks
  Change from baseline to week 4 in Positive and Negative Syndrome Scale (PANSS) total score. Scores range from 23-161; a higher score indicates a more severe illness.
Change in Young Mania Rating Scale (YMRS) total score | 4 weeks
  Change from baseline to week 4 in Young Mania Rating Scale (YMRS) total score. Scores range from 0-60; a higher score indicates a more severe illness.
Change in Extrapyramidal Symptom Rating Scale (ESRS) total score | 4 weeks
  Change from baseline to week 4 in Extrapyramidal Symptom Rating Scale (ESRS) total score. Scores range from 0-102; a higher score indicates more severe symptoms.
Change in Pittsburgh Sleep Quality Index (PSQI) total score | 4 weeks
  Change from baseline to week 4 in Pittsburgh Sleep Quality Index (PSQI) total score. Scores range from 0-21; a higher score indicates worse sleep quality.
Change in Global Functioning Scale - Social and Role (GFS) total score | 4 weeks
  Change from baseline to week 4 in Global Functioning Scale - Social and Role (GFS) total score. Scores range from 6-60; a lower score indicates worse social and role functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Virginie-Anne Chouinard, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States